CLINICAL TRIAL: NCT03456440
Title: The Use of MRI Apparent Diffusion Coefficient Value (ADC Value) to Assess Liver Cirrhosis in Hepatitis C Patients: Observational Case Control Study
Brief Title: The Use of MRI Apparent Diffusion Coefficient Value (ADC Value) to Assess Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jimmy Naaman, principal investigator, Assiut University
Other Study IDs: ADC value and cirrhotic liver
Record Dates: First submitted 2018-02-23; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hepatitis C child pugh's class A: patients are examined with MRI
  Interventions: Diagnostic Test: MRI
- normal individuals: controls cases are examined with MRI
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI scan of the patients liver with DWI and acquisition of ADC value.

SUMMARY:
Hepatitis is known to induce severe liver diseases. The evaluation of the severity of liver cirrhosis is very important for the selection of appropriate treatment plan and the monitoring of patient response to treatment, accurate staging of liver fibrosis is critical because it determines the indication of antiviral treatment and prognosis of patients with chronic viral hepatitis, DWI is a particularly appealing method for the diagnosis of liver fibrosis because it is easy to implement and process, without the need for contrast agents. Apparent diffusion coefficient (ADC) has been shown to be a promising marker of fibrosis and cirrhosis.

DETAILED DESCRIPTION:
Introduction Hepatitis is known to induce severe liver diseases such as liver cirrhosis and liver cancer which are serious threats to public health. The evaluation of the severity of liver cirrhosis is very important for the selection of appropriate treatment plan and the monitoring of patient response to treatment [1].

Noninvasive Child-Pugh classification is a common method to assess liver function, treatment outcome and prognosis in patients with chronic liver cirrhosis [2].

Accurate staging of liver fibrosis (commonly determined by liver biopsy) is critical because it determines the indication of antiviral treatment and prognosis of patients with chronic viral hepatitis. For example, patients with cirrhosis are at higher risk of end-stage liver disease, portal hypertension, and hepatocellular carcinoma and are less likely to respond to antiviral therapy [8-9].

However, liver biopsy is relatively invasive, limited by sample size, and difficult to repeat. Thus, noninvasive tools to assess the degree of fibrosis of the whole liver are urgently needed. Several noninvasive MRI techniques have been investigated for the diagnosis of liver fibrosis and cirrhosis, including diffusion weighted imaging (DWI) [20-24], MR Elastography [25], and perfusion-weighted imaging [26-27].

DWI is a particularly appealing method for the diagnosis of liver fibrosis because it is easy to implement and process, without the need for contrast agents. Apparent diffusion coefficient (ADC) has been shown to be a promising marker of fibrosis and cirrhosis by several independent investigators [20-24].

Recently magnetic resonance Diffusion Weighted Imaging (DWI) has become another noninvasive approach to assess liver cirrhosis by analyzing the changes of water diffusion based on the apparent diffusion coefficient (ADC) [3].

Several studies showed that ADC values of cirrhotic liver were correlated with the results of Child-Pugh classification for the evaluation of the severity of liver cirrhosis [4-7].

However, whether ADC values of cirrhotic liver are correlated with the results of Child-Pugh classification, it remains unclear. The DWI is a specific MRI technique that evaluates the motion of, mainly, water protons in the tissue. The apparent diffusion coefficient (ADC) is the most frequently used DWI measure and provides useful information about inflammation, perfusion and local cell breakdown. The ADC map is calculated based on exponential fitting of DWI over multiple b-values and is used to measure diffusion quantitatively. Prior studies have shown that in liver fibrosis water diffusion may be diminished by extracellular collagen fibers and proteoglycans, thus, reduced ADC values have been reported for liver fibrosis. [10,11,12,13,14,15,16,17,18,20].

These findings suggest DWI could be a useful imaging technique to evaluate fibrosis. In more recent studies, researchers examined the relationship between the stages of hepatic fibrosis and ADC values [14,15,16,19,20].

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C positive patients with Child-Pugh (A) classification.

Exclusion Criteria:

* Advanced liver cirrhosis with decompensated liver or patients with malignant hepatic focal lesions.
* Cases with proven structural abnormalities, history of liver disease or risk factors of liver disease will be excluded from healthy controls.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from outpatient clinic of radiology department of Assiut university hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
changes of MRI ADC value to assess early liver cirrhosis. | 30 minutes
  Hepatitis C patients With child pugh's classification A as Assessed by MRI ADC value changes.

CONTACTS AND LOCATIONS:
Overall Officials: sherif abd elal, MD, Study Director — Assiut university lecturer